CLINICAL TRIAL: NCT03831438
Title: A Phase 1 Open-Label Study to Determine the Safety and Tolerability of AVID200: A Transforming Growth Factor β (TGFβ) Inhibitor, in Patients With Diffuse Cutaneous Systemic Sclerosis
Brief Title: Safety and Tolerability Study of AVID200 in Pts With Diffuse Cutaneous Systemic Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVID200-01
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Scleroderma, Diffuse
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Intervention Model Description: Open-label, uncontrolled, non-randomized study, escalating doses of study drug in sequential patient cohorts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Other): Sequential escalating doses of AVID200 when administered once every 2 weeks (Q2W) by 1-hour intravenous (IV) infusion to patient cohorts with diffuse cutaneous systemic sclerosis (dcSSc).
  Each 2-week dosing period equals 1 cycle; patients may receive up to 3 cycles of AVID200 (i.e., dosing on D1, 15, and 29 of overall 6 week treatment period).
  Interventions: Drug: AVID200

INTERVENTIONS:
Drug: AVID200 — Intravenous infusion of AVID200 Q2 weeks for 3 doses
  Other Names: AVID200 DP

SUMMARY:
Several lines of evidence place TGF-β, a potent pro-fibrotic cytokine, at the centre of the pathogenesis of Systemic Sclerosis (SSC). AVID200 is a novel inhibitor of TGF-β ligands. This Phase 1 trial is designed to evaluate the safety, tolerability and preliminary efficacy of AVID200 in SSc patients in order delineate doses to be further evaluated in Phase 2. Approximately 9 to 24 male and female patients with documented SSc (i.e., score ≥ 9 according to the American College of Rheumatology/European League Against Rheumatism classification criteria), and classified as having the diffuse cutaneous SSs (dcSSc) subset (i.e., according to the LeRoy and Medsger Classification), will be entered into this Phase 1a, multicentre, open-label, dose-escalation, cohort study of AVID200.

DETAILED DESCRIPTION:
The trial is designed to evaluate the safety and tolerability of sequential escalating doses of AVID200 (study drug), in order delineate a potential effective range of tolerated doses to be further evaluated in Phase 2.

Patients will be treated and followed on an outpatient basis throughout the trial, unless hospitalization is required for other reasons, or to assure patient safety. The choice of doses for further Phase 2 study will be based on clinical and laboratory data obtained during this trial, including safety, PK, and preliminary anti-fibrotic activity.

Upon completion of Cycle 1, and provided re-treatment criteria are met, patients may receive up to 2 additional cycles of study drug unless a criterion for treatment discontinuation has been met.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the ability to understand and give written informed consent
* Male or female patients, ≥ 18 years
* Patients classified as having systemic sclerosis (SSc) with a total ≥ 9 according to the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) criteria for the classification of SSc
* Patients classified as having diffuse cutaneous SSc (dcSSc) subset
* Patients with < 5 years since the onset of first SSc manifestations, other than Raynaud's phenomenon, at the time of enrollment
* Patients with a MRSS ≥ 15, and with a score that has not decreased by > 5 points in the past 2 months (8 weeks)
* Patients with a skin score ≥ 2 on at least one forearm
* Persons of childbearing potential agreeing to use a highly effective, non-hormonal method of contraception during the study

Exclusion Criteria:

* Women who are pregnant or intending to become pregnant before study, during study or within 3 months after the last dose of study drug; women who are breastfeeding
* Patients with any of the following hematologic abnormalities at baseline:

  * Hemoglobin < 10.0 g/dL*
  * Absolute neutrophil count (ANC) < 1,500 per mm3
  * Platelet count < 100,000 per mm3
  * Iron, iron binding, and transferrin studies to be performed at screening; patients with documented iron deficiency to receive repletion prior to receiving study drug
* Patients with any of the following serum chemistry abnormalities at baseline:

  * Total bilirubin ≥ 1.5 × the ULN for the institution
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 2.5 × the ULN for the institution (≥ 5× ULN if due to hepatic involvement by disease)
* History of scleroderma renal crisis within 6 months or creatinine > 2.0 mg/dL
* Lack of intravenous (IV) access required for study drug administration
* History of organ transplantation (e.g., stem cell or solid organ)
* Patients with:Active uncontrolled bleeding or a known bleeding diathesis, Active thrombosis, thrombophlebitis, thromboembolism, or hypercoagulable state
* Patients with a significant cardiovascular disease or condition, including:

  * Congestive heart failure (CHF), Left ventricular ejection fraction (LVEF) known to be below the lower limit of normal (LLN) for the center, or < 50% by multi-gated acquisition (MUGA) scan or echocardiogram (ECHO) if no LLN is defined by the site
* Need for antiarrhythmic medical therapy for a significant ventricular arrhythmia or other uncontrolled arrhythmia
* Severe conduction disturbance (i.e., trifascicular heart block)
* QTc interval ≥ 480 msec
* Uncontrolled hypertension (per the Investigator's discretion)
* History of acute coronary disease (including myocardial infarction [MI] and angina), coronary angioplasty, stenting, or bypass surgery within 2 years
* Patients with a significant pulmonary disease or condition
* History of ascites or pleural effusion, unless successfully treated and completely resolved and the patient has not been treated for the conditions for > 4 months prior to first study drug administration
* Significant gastrointestinal (GI) or hepatic disease or condition, including but not limited to:
* GI involvement requiring total parenteral nutrition or hospitalization for pseudo-obstruction within 3 months prior to first study drug administration
* Moderate to severe hepatic impairment (i.e., Child-Pugh Class B or C)
* Patients with an active malignancy or history of a malignancy within the last 2 years with specified exceptions
* Patients with a known or suspected hypersensitivity to any of the excipients of formulated AVID200
* Patients with any of the following, Human immunodeficiency virus (HIV) infection (i.e., HIV RNA-positive)
* Active/chronic infection with hepatitis B virus (HBV) (i.e., HB surface antigen [HBsAg]-positive, HB surface antibody [HBsAb]-negative)
* Active/chronic infection with hepatitis C virus (HCV) (i.e., HCV RNA-positive)
* Patients with known active bacterial, viral, fungal, mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of the nail bed), or any other serious/active/uncontrolled infection, any infection requiring hospitalization or treatment with parenteral antibiotics, or unexplained fever > 38.5ºC within 4 weeks prior to first study drug administration
* Patients with unresolved > Grade 1 adverse event (AE) associated with any prior therapy for dcSSc
* Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure within 4 weeks prior to first study drug administration
* Patients with any other serious, life-threatening, or unstable preexisting medical condition (aside from the underlying diagnosis), including significant organ system dysfunction, or clinically significant laboratory abnormality (ies), which, in the opinion of the Investigator, would either compromise the patient's safety, significantly increase the risk of SAEs, limit life expectancy, or interfere with obtaining informed consent, compliance with study procedures, or evaluation of the safety of the study drug
* Patients with ongoing drug or alcohol abuse that would impact compliance with study-related procedures or evaluations
* Patients with a psychiatric disorder, or altered mental status that would preclude understanding of the informed consent process and/or completion of the necessary study-related evaluations
* Patients with the inability or with foreseeable incapacity, in the opinion of the Investigator, to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Incidence of treatment related adverse events | 10 Months
  Incidence of treatment related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lafyatis, MD, Study Chair — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Hospital of Special Surgery, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania